CLINICAL TRIAL: NCT05958823
Title: Evaluation of the Effects of Serratus Anterior Plan Block (SAP) and Pectoralis Blocks (PECS I-II) on the Postoperative Period After Open Heart Surgery
Brief Title: Effects of Serratus Anterior Plan Block (SAP) and Pectoralis Blocks (PECS I-II) After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 22.05.2023-1
Record Dates: First submitted 2023-05-23; First posted 2023-07-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Pain; Postoperative Complications; Side Effect
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: randomized, controlled, prospective
Who Masked: Participant, Care Provider
Masking Description: Results evaluators and surgeons will be unaware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Serratus anterior plane block) (Experimental): The patient who underwent open heart surgery will be taken to the cardiovascular surgery intensive care unit after the surgical procedure. Necessary preparations will be made to perform serratus anterior plane block (SAP). After ensuring the hygiene of the anterior chest wall, it is advanced with an 8 cm long peripheral block needle under ultrasound guidance. SAP block is a local anesthetic injection procedure applied superficially or deeply to the serratus anterior muscle and specifically targeting the lateral cutaneous and muscular branches of the intercostal nerves. The long thoracic nerve and the thoracodorsal nerve are located in the fascial plane on the surface of the serratus anterior muscle and can be blocked. The serratus anterior block can be performed anywhere between the anterior and posterior axillary lines and the 2nd and 7th ribs.
  Interventions: Procedure: Serratus anterior plane block
- Group P ( PECS I-II) (Experimental): The patient who underwent open heart surgery will be taken to the postoperative intensive care unit. Preparation for the PECS block will be made, and after the anterior chest wall hygiene is ensured, an 8 cm long peripheral block needle will be advanced under ultrasound guidance. PECS II block is a combination of PECS I and subpectoral local anesthetic injection targeting the lateral cutaneous branches of the intercostal nerves, long thoracic and thoracodorsal nerves. To perform the PECS I block, the ultrasound probe is placed in the midclavicular line and in the parasagittal plane, and the pectoralis major-minor, axillary vessels and pleura are visualized. After identifying the second and third ribs by sliding the ultrasound probe caudally, the lower end will be rotated towards the axilla to make the probe parallel to the deltapectoral groove.
  Interventions: Procedure: PECS I-II

INTERVENTIONS:
Procedure: Serratus anterior plane block — Serratus anterior plane block
  Arms: Group S (Serratus anterior plane block)
Procedure: PECS I-II — PECS I-II
  Arms: Group P ( PECS I-II)

SUMMARY:
The effects of anterior chest wall blocks (PECS and SAP will be used in this study) performed for postoperative analgesia on pain scores (to be checked with visual analogue scale (VAS), opioid consumption, length of hospital stay, mobilization time, side effects and complications in the postoperative period will be examined.

DETAILED DESCRIPTION:
Patients who were taken in accordance with the inclusion criteria and signed the consent form will be randomly divided into 2 groups. Randomization: Patients will be randomly divided into 2 groups using the closed envelope method:

Group S (Those who will have serratus anterior plane block): The patient who has undergone coronary bypass surgery will be taken to the cardiovascular intensive care unit after the surgical procedure. Necessary preparations will be made to make an SAP block. After ensuring the hygiene of the anterior chest wall, it is advanced with an 8 cm long peripheral block needle under ultrasound guidance. SAP block is a local anesthetic injection procedure applied superficially or deeply to the serratus anterior muscle and specifically targeting the lateral cutaneous and muscular branches of the intercostal nerves. The long thoracic nerve and the thoracodorsal nerve are located in the fascial plane on the surface of the serratus anterior muscle and can be blocked. The serratus anterior block can be performed anywhere between the anterior and posterior axillary lines and the 2nd and 7th ribs. It is performed with the patient in the supine position with the ipsilateral arm abducted 90 degrees or in the lateral decubitus position with the operative side up, while the same side arm is flexed and extended forward. The SAP block will be performed at the level of the 4th rib. The injection site will be found by placing the ultrasound probe under the clavicle in a parasagittal manner and counting from the second rib. By moving the probe laterally towards the mid or posterior axillary line, the serratus anterior muscle will be seen as a layer of muscle over the anechoic shadow of the rib. It extends over the latissimus dorsi serratus anterior muscle and will appear thicker and more prominent in the posterior axillary line. The needle will be advanced superficially or deep to the serratus anterior muscle and 30 mL of local anesthetic (bupivacaine) will be administered to the fascial plane.

Group P (PECS I-II): The patient who has undergone coronary bypass surgery will be taken to the postoperative intensive care unit. Preparation for the PECS block will be made, and after the anterior chest wall hygiene is ensured, an 8 cm long peripheral block needle will be advanced under ultrasound guidance. PECS II block is a combination of PECS I and subpectoral local anesthetic injection targeting the lateral cutaneous branches of the intercostal nerves, long thoracic and thoracodorsal nerves. To perform the PECS I block, the ultrasound probe is placed in the midclavicular line and in the parasagittal plane, and the pectoralis major-minor, axillary vessels and pleura are visualized. After identifying the second and third ribs by sliding the ultrasound probe caudally, the lower end will be rotated towards the axilla to make the probe parallel to the deltopectoral groove. Combined with the in-plane technique, this rotation provides better extension to the intercostobrachial nerve. The tip of the needle will be placed in the interpectoral fascial plane (between pectoralis major and minor) and 15 mL of local anesthetic (bupivacaine) will be injected. To perform the PECS II block, in addition to the PECS I block, the needle is advanced from the interpectoral fascial plane to the fascial plane between the pectoralis minor and the serratus anterior. 15mL or local anesthetic (bupivacaine) will be injected into this area (for 15 ml PECS I, a total of 30ml local anesthetic for 15 ml PECS II). An investigator not associated with the study will perform randomization using a computer generated randomization table.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study,
* 20-65 years old
* ASA I-II-III
* Open heart surgery

Exclusion Criteria:

* Refusal to participate in the study
* 20 years old, over 65 years old
* Pregnancy
* Presence of bleeding diathesis
* Liver or kidney failure
* Receiving effective treatment on immunity
* Immune suppressed
* Those with BMI ≥30

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia | postoperative 24 hour
  will be evaluated with VAS (vsual anlague scale) VAS 0-2: no pain, 3-4: mild pain, 5-6: moderate pain, 7-8: severe pain, 9-10: excruciating pain

SECONDARY OUTCOMES:
side effects | postoperative 4.hour(only once)
  nausea, vomiting will be observed
complications | postoperative 24 hour
  ultrasonography will be used to minimalized complications

CONTACTS AND LOCATIONS:
Overall Officials: School of Medicine Department of Anesthesiology and Reanimation, Study Chair — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
participiants's personal information will not be shared anyone